CLINICAL TRIAL: NCT02432664
Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of Single and Multiple Escalating Doses of ODM-108: A Single Centre Study in Healthy Male Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Effects of ODM-108: in Healthy Male Volunteers
Acronym: FIMTRIP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated after the second cohort had completed Part II due complex PK results. There were no safety concerns.
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3118001
Record Dates: First submitted 2015-04-02; First posted 2015-05-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ODM-108 Part I (Experimental): Oral capsules dosage 0.2 - 240 mg once daily for one day
  Interventions: Drug: ODM-108 Part I
- Placebo Part I (Placebo Comparator): Oral capsules given once daily for one day
  Interventions: Drug: Placebo Part I
- ODM-108 Part II (Experimental): Oral capsules 4 dose levels to be decided after Part 1 of the study. 1 - 4 times a day for 7 days
  Interventions: Drug: ODM-108-Part II
- Placebo Part II (Placebo Comparator): Oral capsules 1 - 4 times per day for 7 days
  Interventions: Drug: Placebo Part II
- ODM-108 Part III (Experimental): Oral capsules 1-4 times daily for 7 to 10 days
  Interventions: Drug: ODM-108 Part III
- Midazolam (Active Comparator): Single dose as a solution 3 days prior to the first dose of ODM-108 and on the last day of dosing with ODM-108
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: ODM-108 Part I — Single oral escalating dose of ODM-108. Each volunteer will receive either one dose of ODM-108 or placebo
  Arms: ODM-108 Part I
Drug: Placebo Part I — Single oral escalating dose of ODM-108. Each volunteer will receive either one dose of ODM-108 or placebo
  Arms: Placebo Part I
Drug: ODM-108-Part II — Multiple escalating doses based on the results of Part 1. Either ODM-108 or placebo 1 - 4 times a day for 7 days
  Arms: ODM-108 Part II
Drug: Placebo Part II — Multiple escalating doses based on the results of Part 1. Either ODM-108 or placebo 1 - 4 times a day for 7 days
  Arms: Placebo Part II
Drug: ODM-108 Part III — Oral capsules 1 - 4 times daily for 7 to 10 days
  Arms: ODM-108 Part III
Drug: Midazolam — Single dose as a solution 3 days prior to the first dose of ODM-108 and on the last day of dosing with ODM-108
  Arms: Midazolam

SUMMARY:
The purpose of the study is to investigate to what extent this new study drug is tolerated in humans.

The study is divided into 3 parts (Part III is optional and may go ahead depending on the results of Parts I and II). The volunteers will only be enrolled to one part of the study. In parts I and II the volunteer will receive active study drug or placebo. In part I the volunteers will receive a single dose of one of the eight planned escalating dose levels.

In part II volunteers will receive 4 planned dose levels based on the results obtained in Part 1 of the study, with the option to include an additional dosing group.

In optional part III the volunteer will receive ODM-108 and an already registered drug so that interactions with other drugs can be studied.

It will be investigated how quickly and to what extent the study drug is absorbed and eliminated from the body (this is called pharmacokinetics). In addition, in parts I and II the effect of the compound on the sensation of pain and on cognition (activities of thinking, understanding, learning, and remembering) will be investigated (this is called pharmacodynamics).

DETAILED DESCRIPTION:
This is the first time that this compound is being given to humans.

The study will only take place after it has been approved by the Independent Ethics Committee.

ELIGIBILITY:
Inclusion Criteria applicable to Parts I - III:

* Written informed consent.
* Good general health
* Males between 18 and 55 years (inclusive).
* Body mass index (BMI) between 18-30 kg/m2 inclusive
* Weight 55-95 kg (inclusive).
* Participants with female partners of child-bearing potential must adhere to a proper form of contraception.
* Subjects with light coloured skin.

Exclusion Criteria:

* A predictable poor compliance or inability to understand and comply with the protocol , instructions and protocol restrictions or communicate well with the investigator.
* Vulnerable subjects.
* Veins unsuitable for repeated venipuncture.
* Evidence of clinically relevant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
* Medical history of relevant psychiatric disorders or evidence of clinically relevant neuropsychiatric disease.
* Suicidal ideation in the 6 months before screening or current risk of suicide based on the investigators judgement.
* History of hypersensitivity to drugs or excipients.
* Any condition requiring regular concomitant medication.
* Intake of any medication that could affect the outcome of the study.
* History of Alcoholism.
* Inability to refrain from using nicotine-containing products for 48 h before and during the stay in the study centre.
* History of drug abuse or positive drug screen.
* Blood donation or loss of a clinically relevant amount of blood within 2 months before the screening visit.
* Abnormal 12-lead ECG
* Heart rate < 40 bpm or > 100 bpm at screening.
* Systolic BP < 90 mmHg or > 140 mmHg, diastolic BP< 45 mmHg or > 90 mmHg, orthostatic hypotension - decrease of more than or equal to 20 mmHg for systolic BP, decrease of more than or equal to 10 mmHg for diastolic BP at screening.
* Abnormal 24-h Holter of clinical relevance at screening.
* Positive serology for HIV antibodies (HIVAb), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCVAb).
* Thrombocytes and neutrophils count is < the lower limit of normal range.
* alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase and total bilirubin > upper limit of normal (ULN).
* Any abnormal value of laboratory, vital signs, or physical examination, which may, in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk for the subject.
* Participation in an investigational drug study within 2 months before entry into this study.
* An employee or direct relative of the employee of the CRO or sponsor.
* Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk for the subject.

Additional exclusion criteria for Part I and II:

* An abnormal screening EEG.
* A history of skin conditions or bad reactions after exposure to capsaicin or mustard oil.
* Following intradermal injection of capsaicin (100 μg) at screening visit, the area of hyperalgesia was < 10 cm2, or if the area of flare < 10 cm2 at 15 min.

Additional exclusion criterion for Part II:

* Use of nicotine-containing products within the previous 3 months.

The following additional exclusion criterion will be checked in Part I and II:

* Inability to complete either Digital Symbol Substitution Test (DSST) (for Part I) or psychomotor test battery (for Part II).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events in Part I and Part II. | From screening up to 8 weeks
  Clinically relevant changes from baseline of safety assessment

SECONDARY OUTCOMES:
Part III (optional) Effect of ODM-108 on the activity of CYP3A4 (cytochrome P450 3A4) isoenzymes | Day 1 up to Day 11
  Measurement of biomarkers
Part I Peak plasma concentration Cmax of ODM-108 | Pre dose,15, 30, 45 mins, 1 h, 1 h 15, 1 h 30, 2 h, 2 h 30, 3 h, 4 h, 6 h, 8 h, 12h, 24 h, 48 h, 72 h, 96 h post dose at each dose level.
  Cmax of ODM-108 after single dosing
Part I Metabolite screening in plasma and urine | Pre-dose and 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h and 48 h post dose at each dose level. Urine samples pre-dose and for 24 hours post dose at each dose level.
  Metabolite screening in plasma and urine after single dosing
Part I Sedation scores on Visual Analogue Scales | Pre-dose, 2 h 30 min and 10 h post dose at each dose level
  Assessment of sedation by subject
Part I Cognitive function - Digital Symbol Substitution Test | Pre-dose, 2 h 30 min and 10 h post dose at each dose level
  Assessment of cognitive function
Part I Intensity of spontaneous pain | Screening and day 1 at 1, 5, 15, 30, 60 and 120 min after capsaicin injection.
  Intensity of spontaneous pain as assessed by a visual analogue scale
Part I Area of hyperalgesia | Screening and day 1 at 15, 30, 60 and 120 min after capsaicin injection.
  Area of hyperalgesia quantified by a Von Frey monofilament
Part I area of flare response | Screening and day 1 at baseline and 15, 30, 60 and 120 min after capsaicin injection.
  Area of flare response measured by Doppler blood flow scan
Part II Peak plasma concentration Cmax of ODM-108 | Days 1 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  Cmax of ODM-108 after multiple dosing
Part II Peak plasma concentration Cmax of ODM-108 fed day 5 period 1 | Days 1,5 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  Cmax of ODM-108 after multiple dosing
Part II Time to peak plasma concentration (tmax) of ODM-108 | Days 1 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  tmax of ODM-108 after multiple dosing
Part II Time to peak plasma concentration (tmax) of ODM-108 fed day 5 period 1 | Days 1,5 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  tmax of ODM-108 after multiple dosing
Part II Area under the plasma concentration versus time curve (AUC) of ODM-108. | Days 1 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  AUC of ODM-108 after multiple dosing
Part II Area under the plasma concentration versus time curve (AUC) of ODM-108 fed day 5 period 1 | Days 1,5 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  AUC of ODM-108 after multiple dosing
Part II Elimination half-life of ODM-108 | Days 1 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  Elimination half-life of ODM-108 after multiple dosing
Part II Elimination half-life of ODM-108- fed day 5 period 1 | Days 1,5 and 7: Pre-dose and 0.25, 0.5, 0.75,1,1.25,1.5, 2, 2.5, 3,4,6,8,12h post dose. Day 2-6 pre-dose, Day 7: 24, 48, 72 and 96h post dose
  Elimination half-life of ODM-108 after multiple dosing
Part II Binding of ODM-108 to proteins in plasma | Days 1 and 7 -1 h 30 min post dose
  Assessment of binding of ODM-108 to proteins in plasma
Part II Metabolite screening in plasma and urine | Day 1 and 7 pre-dose and 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h and 48 h post dose. Urine samples pre-dose and for 24 hours post dose at each dose level on days 1 and 7.
  Metabolite screening in plasma and urine
Part II Sedation scores on Visual Analogue Scales | Day 1 and day 6 pre-dose, 2 h 30 min, and 10 h post dose
  Assessment of sedation by subject
Part II Computerised psychomotor test battery measuring: attention, concentration, vigilance, memory, visual motor coordination and body sway. | Days 1 and 6: pre-dose, approx. 2 h 30 min and 10 h after first daily ODM-108 dose
  Assessment of psychomotor function
Part II Intensity of spontaneous pain | Screening and day 5 at 1, 5, 15, 30, 60 and 120 min after capsaicin injection.
  Assessed by numerical rating scale
Part II Area of hyperalgesia | Screening and day 5 at 5, 15, 30, 60 and 120 min after capsaicin injection.
  Area of hyperalgesia quantified by a Von Frey monofilament
Part II Cutaneous blood flow and area of flare response | Screening and day 5 pre -dose and 5, 15, 30, 60 and 120 min after capsaicin injection.
  Pain assessments
Part II Intensity of spontaneous pain | Screening and day 7 at 1, 5, 15, 30, 60 and 120 min after mustard oil challenge.
  Intensity of spontaneous pain as assessed by a visual analogue scale
Part II Area of hyperalgesia | Screening and day 7 at 5, 15, 30, 60 and 120 min after mustard oil challenge.
  Area of hyperalgesia quantified by a Von Frey monofilament
Part II Area of flare response | Screening and day 7 baseline and 5, 15, 30, 60 and 120 min after mustard oil challenge.
  Area of flare response measured by Doppler blood flow scan
Part III (optional) Peak plasma concentration Cmax of midazolam | day 1 and day 10 or 13
  Cmax of midazolam
Part III (optional) Time to peak plasma concentration (tmax) of midazolam | day 1 and day 10 or 13
  tmax of midazolam
Part III (optional) Area under the plasma concentration versus time curve (AUC) of midazolam. | day 1 and day 10 or 13 (
  AUC of midazolam
Part III (optional) ODM-108 levels in cerebrospinal fluid | day 9
  Assessment of levels of ODM 108 in cerebrospinal fluid
Part I Time to peak plasma concentration (tmax) of ODM-108 | Pre dose,15, 30, 45 mins, 1 h, 1 h 15,1 h 30, 2 h, 2 h 30, 3 h, 4 h, 6 h, 8 h, 12h, 24 h, 48 h, 72 h, 96 h post dose at each dose level.
  tmax of ODM-108 after single dosing
Part I Area under the plasma concentration versus time curve (AUC) of ODM-108. | Pre dose,15, 30, 45 mins, 1 h, 1 h 15,1 h 30, 2 h, 2 h 30, 3 h, 4 h, 6 h, 8 h, 12h, 24 h, 48 h, 72 h, 96 h post dose at each dose level.
  AUC of ODM-108 after single dosing
Part I Elimination half-life of ODM-108 | Pre dose,15, 30, 45 mins, 1 h, 1 h 15,1 h 30, 2 h, 2 h 30, 3 h, 4 h, 6 h, 8 h, 12h, 24 h, 48 h, 72 h, 96 h post dose at each dose level.
  Elimination half-life of ODM-108 after single dosing

CONTACTS AND LOCATIONS:
Overall Officials: Sjoerd van Marle, M.D, Principal Investigator — PRA Health Sciences; Sara Haworth, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- PRA Health Sciences, Zuidlaren, Netherlands